CLINICAL TRIAL: NCT00660881
Title: A Phase IIb Multi-Center, Open-label, Follow-up Study to Assess Safety and Efficacy of Epratuzumab in Serologically-positive Systemic Lupus Erythematosus Patients With Active Disease Who Participated in Study SL0007
Brief Title: Open-label Study of Epratuzumab in Serologically-positive Systemic Lupus Erythematosus Patients With Active Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL0008; EudraCT Number: 2007-002589-37
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Monoclonal antibody; B-Cell immunotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EMAB (Experimental): 1200 mg epratuzumab given in 2 doses every other week in 12 week treatment cycles.
  Interventions: Biological: Epratuzumab

INTERVENTIONS:
Biological: Epratuzumab — Epratuzumab at a concentration of 10 mg/mL prepared in 17.5 ml vials for slow intravenous infusion using only PBS as a vehicle/buffer for the infusion procedure.

SUMMARY:
The primary objective of the study is to assess the safety of epratuzumab in patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

* SL0007 patients who completed through week 12 of the study or who early terminated at week 8 or later due to treatment failure
* Patients must have maintained eligibility requirements throughout their participation in SL0007
* Written informed consent signed prior to initiation of any study-specific assessments at visit 1

Exclusion Criteria:

* Patients may not receive any live vaccination within 2 weeks prior to visit 1 or during the course of the study
* Active severe SLE disease activity which involves the CNS system (defined by BILAG neurologic A level activity) including transverse myelitis, psychosis and seizures
* Active severe SLE disease activity which involves the Renal system (defined by BILAG renal level A activity or Grade III or higher WHO nephritis) or serum creatinine >2.5mg/dL or clinically significant serum creatinine increase within the prior 4 weeks or proteinuria >3.5gm/day
* Patients with a history of anti-phospholipid antibody syndrome AND Use of oral anticoagulants or anti-platelet treatment
* Patients with a history of chronic infection, recent significant infection, or any current sign of symptom that may indicate an infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Continue to assess safety of epratuzumab by assessing adverse events (including infusion reactions), vital signs and clinical safety laboratory assessments (Timeframe: All visits) | 12 Week treatment cycles

SECONDARY OUTCOMES:
The combined response index analysis evaluating BILAG, SLEDAI, and a physician's global assessment and treatment failure status | Every 4 weeks through week 48, then every 12 weeks through completion
The combined response index including an additional criteria involving the SF-36 response | Every 12 weeks
BILAG score assessment | Every 4 weeks through week 48, then every 12 weeks through completion
SLEDAI scores assessment | Every 4 weeks through week 48, then every 12 weeks through completion
Patient and physician VAS | Every 4 weeks through week 48, then every 12 weeks through completion
Percentage of patients achieving SF-36 stabilization or improvement as compared to baseline | Every 12 weeks
SF-36 PCS, MCS | Every 12 weeks
EQ-5D results | Every 12 weeks
Proportion of patients meeting treatment failure | Every 12 weeks
Total daily steroid dose | Every 4 weeks for the first 48 weeks and then every 12 weeks
Time to flare for patients who entered the study without flare as defined by the BILAG | over the entire course of the trial
SLEDAI responder | Every 4 weeks for the first 48 weeks and then every 12 weeks
Time to sustained response for patients entering SL0008 with flare as defined by the BILAG. | over the entire course of the trial
Immunogenicity as measured by human anti-human antibodies | at each dosing visit and 4 weeks post first dose of each treatment cycle
Assessment of changes in baseline in levels of circulating B and T cells | The first dosing visit of each treatment cycle and at 4 weeks post first dose of each treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (42):
- United States (14):
  - Birmingham, Alabama
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - San Leandro, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Tampa, Florida
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Wilmington, North Carolina
  - Oklahoma City, Oklahoma
  - Arlington, Virginia
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (3):
  - Goiânia, Goiás
  - Porto Alegre
  - São Paulo
- Shatin, Hong Kong
- Hungary (2):
  - Debrecen
  - Zalaegerszeg
- India (5):
  - Madurai, Tamil Nadu
  - Bangalore
  - Hyderabad
  - Manipal
  - Nagpur
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (5):
  - Elblag
  - Gmina Końskie
  - Lublin
  - Poznan
  - Torun
- Spain (2):
  - Barcelona
  - Santander
- Ukraine (4):
  - Donetsk
  - Ivano-Frankivsk
  - Kiev
  - Lviv
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Wallace DJ, Hobbs K, Clowse ME, Petri M, Strand V, Pike M, Merrill JT, Leszczynski P, Neuwelt CM, Jeka S, Houssiau F, Keiserman M, Ordi-Ros J, Bongardt S, Kilgallen B, Galateanu C, Kalunian K, Furie R, Gordon C. Long-Term Safety and Efficacy of Epratuzumab in the Treatment of Moderate-to- Severe Systemic Lupus Erythematosus: Results From an Open-Label Extension Study. Arthritis Care Res (Hoboken). 2016 Apr;68(4):534-43. doi: 10.1002/acr.22694. PMID 26316325